CLINICAL TRIAL: NCT06300151
Title: The Effect of Ultrasound Real-time Guidance Technique on the Effectiveness and Safety of Labor Analgesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zongxun Lin (Other)
Responsible Party: Sponsor-Investigator, Zongxun Lin, Principal Investigator, Fujian Provincial Hospital
Organization: Fujian Provincial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ultrasound Real-time Guidance
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Labor Analgesia
Keywords: Ultrasound Real-time Guidance; labor analgesia; delivery woman; neonate; Effectiveness; Safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound Real-time Guidance combined with Dural Puncture Epidural Group (Experimental): Ultrasound real-time guidance combined with dural puncture epidural Can improve the clinical effect of labor analgesia.
  Interventions: Device: Ultrasound Real-time Guidance combined with Dural Puncture Epidural Labor Analgesia
- Dural Puncture Epidural Group (Active Comparator): Dural Puncture Epidural is a clinical improvement of Combined Spinal-Epidural and is widely used in Maternal. The implementation step is to complete the epidural puncture, temporarily do not place a tube, puncture the dura mater with a subarachnoid anesthesia needle, but do not directly inject drugs into the subarachnoid space, and then leave an epidural catheter for administration according to epidural block.
  Interventions: Device: Dural Puncture Epidural Labor Analgesia

INTERVENTIONS:
Device: Ultrasound Real-time Guidance combined with Dural Puncture Epidural Labor Analgesia — Ultrasound real-time guidance technology has great advantages over traditional blind exploration technology in terms of accuracy, success rate, and reduction of puncture damage in intervertebral space positioning through operational visualization, greatly improving the effectiveness and safety of spinal block.
  Arms: Ultrasound Real-time Guidance combined with Dural Puncture Epidural Group
Device: Dural Puncture Epidural Labor Analgesia — Dural Puncture Epidural is a clinical improvement of Combined Spinal-Epidural and is widely used in Maternal. The implementation step is to complete the epidural puncture, temporarily do not place a tube, puncture the dura mater with a subarachnoid anesthesia needle, but do not directly inject drugs into the subarachnoid space, and then leave an epidural catheter for administration according to epidural block.
  Arms: Dural Puncture Epidural Group

SUMMARY:
Ultrasound real-time guidance technology has great advantages over traditional blind exploration technology in terms of accuracy, success rate, and reduction of puncture damage in intervertebral space positioning through operational visualization, greatly improving the effectiveness and safety of spinal block. At present, Doppler ultrasound is rarely used for spinal block, especially for real-time ultrasound guidance technology, which has not been widely applied in clinical practice due to its high equipment requirements, lack of mature puncture plans, complex operation, and high learning curve. If a comprehensive diagnosis and treatment plan can be developed, it will greatly improve the delivery experience of mothers.

DETAILED DESCRIPTION:
Traditional blind exploration of spinal canal puncture has many limitations, often forcing changes in anesthesia methods due to multiple puncture failures. However, the application of real-time ultrasound guidance technology in spinal canal puncture can completely solve this clinical difficulty. The ultrasound-guided real-time paramedian approach epidural puncture for labor analgesia is a new type of labor analgesia technology, and its specific operating standards and diagnostic and treatment routines have not yet been established, including the selection of puncture path, puncture needle model, distance between puncture hole and epidural injection point, drug type, dosage, solubility, volume and other parameters, all of which have great research space.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) Class I or II;
2. Single healthy pregnancy;
3. Head showing first;
4. 37 to 41 weeks;
5. The labor process is active, and the cervix dilates<5cm;
6. Require epidural labor analgesia;
7. Volunteer to participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Presence of pregnancy diseases, such as pregnancy hypertension, pre eclampsia, pregnancy diabetes;
2. Contraindications to intraspinal analgesia: 1) Central nervous system diseases. 2) Infection or septicemia at the puncture site. 3) Coagulation dysfunction;
3. Known cases of fetal malformation or increased risk of cesarean section, such as a history of uterine rupture;
4. Persons with a history of mental illness, hysteria, epilepsy, etc. who cannot cooperate.
5. Patients with long-term use of opioids, steroids, and chronic pain.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Analgesic effect（onset time） | 7 weeks
  Analgesic effect of pregnant women（onset time）
Analgesic effect（block level） | 7 weeks
  block level of pregnant women by Alcohol swab（temperature sensation：Pubic symphysis=T12，umbilical region=T10，hypochondrium=T8，xiphoid process=T6，Nipple connection=T4，subclavian=T2）
Analgesic effect（block effect） | 7 weeks
  block effect of pregnant women by Alcohol swab（temperature sensation：Unblocked, unilateral block, bilateral block）
Analgesic effect（Visual Analogue Scale） | 7 weeks
  Analgesic effect of pregnant women by Visual Analogue Scale（scale title=Visual Analogue Scale，Total score=0-10,0=no pain,10=worst possible pain）
Analgesic effect（number of Patient controlled analgesia） | 7 weeks
  number of Patient controlled analgesia（Press the PCA button when the patient feels pain）
Analgesic effect（time of Patient controlled analgesia） | 7 weeks
  time of Patient controlled analgesia（Press the PCA button when the patient feels pain）
Uterine contraction indicators（Frequency） | 7 weeks
  Assess uterine contractions（Frequency）
Uterine contraction indicators（duration） | 7 weeks
  Assess uterine contractions（duration）
Uterine contraction indicators（Number of pregnant women with Tachysystole） | 7 weeks
  Tachysystole=More than 5 Uterine contraction in 10 minutes
Uterine contraction indicators（Number of pregnant women with hypertonus） | 7 weeks
  hypertonus=Each Uterine contraction lasts for more than 2 minutes
Fetal heart indicators（Fetal heart rate） | 7 weeks
  Assess fetal heart（Fetal heart rate）
Fetal heart indicators（NICHD classification） | 7 weeks
  Assess fetal heart（NICHD classification）
Fetal heart indicators（Fetal Heart Rate decelerations） | 7 weeks
  Assess fetal heart（Fetal Heart Rate decelerations）
Fetal heart indicators（Fetal Heart Rate Variability） | 7 weeks
  Assess fetal heart（Fetal Heart Rate Variability）
Apgar score | 7 weeks
  Apgar score（scale title=Apgar score，Total score=0-10，0-3=severe asphyxia，4-7=mild asphyxia，8-10=normal）
Sacral sensory block of pregnant women | 7 weeks
  Sacral sensory block of pregnant women by Alcohol swab（temperature sensation：Unblocked, unilateral block, bilateral block）
modified bromage score | 7 weeks
  modified bromage score（scale title=modified bromage score，Total score=0-3，0=no Motor nerve block; 1=unable to lift straight legs, but able to bend knees and move feet; 2=unable to lift straight legs or bend knees, but able to move feet; 3=unable to bend ankles, feet, or knees (completely blocked)）

SECONDARY OUTCOMES:
Operation evaluation（Time） | 7 weeks
  Assessment of puncture condition（Time）
Operation evaluation（number of times） | 7 weeks
  Assessment of puncture condition（number of times）
Operation evaluation（side effects and Complications） | 7 weeks
  Assessment of puncture condition（side effects and Complications）
Delivery mode | 7 weeks
  natural labor/cesarean section/instrument
Concentration of Interleukin 6 | 7 weeks
  Pregnant women's venous blood Interleukin 6
Concentration of hypersensitive C-reactive protein | 7 weeks
  Pregnant women's venous blood hypersensitive C-reactive protein
Concentration of cortisol | 7 weeks
  Pregnant women's venous blood cortisol
Maternal rehabilitation indicators（Postpartum hospital stay） | 7 weeks
  Postpartum hospitalization days
Maternal rehabilitation indicators（Edinburgh Postnatal Depression Scale） | 7 weeks
  Edinburgh Postnatal Depression Scale（scale title=Edinburgh Postnatal Depression Scale，Total score=0-30，≥13=Postpartum depression）
Maternal rehabilitation indicators（Postoperative Recovery Quality Scale（QOR-40）） | 7 weeks
  Postoperative Recovery Quality Scale（QOR-40）（scale title=Postoperative Recovery Quality Scale（QOR-40），Total score=0-200，The higher the score the better the recovery）
Number of pregnant women with adjust the treatment plan and adjustment method | 7 weeks
  adjustment method include Adjust the Epidural catheter or Adjusting drug dosage
Drug consumption | 7 weeks
  Drug consumption
Effect of stages of labor（time） | 7 weeks
  Effect of stages of labor（time）
body temperature changes | 7 weeks
  body temperature changes
Number of pregnant women with Infection during labor | 7 weeks
  whether Infection during labor of pregnant women
Side effects and complications of labor analgesia | 7 weeks
  Side effects and complications of labor analgesia
The reasons and number of pregnant women with conversion of natural labor to Caesarean section | 7 weeks
  Reasons and number for conversion of natural labor to Caesarean section (pregnant woman, fetus, anesthesia, others)
Self-Rating Anxiety Scale | 7 weeks
  Self-Rating Anxiety Scale（scale title=Self-Rating Anxiety Scale，Total score=0-80，≥50=Anxiety）
Delivery fear score（numerical rating scale） | 7 weeks
  Delivery fear score by numerical rating scale（scale title=numerical rating scale，Total score=0-10，≥6=Delivery fear）
Delivery satisfaction survey | 7 weeks
  Delivery satisfaction survey(0=very satisfied, 1=satisfied, 2=common, 3=dissatisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Zongxun Lin, Master, Principal Investigator — Fujian Provincial Hospital
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No